CLINICAL TRIAL: NCT04092270
Title: A Phase I/Ib Dose Escalation Study of Pegylated Liposomal Doxorubicin (PLD) With Peposertib (M3814) in Platinum - Resistant or Ineligible Ovarian and Related Cancers With Planned Expansions in High Grade Serous (HGSOC) and Low Grade Serous Ovarian Cancer (LGSOC)
Brief Title: A Study Combining the Peposertib (M3814) Pill With Standard Chemotherapy in Patients With Ovarian Cancer With an Expansion in High Grade Serous Ovarian Cancer and Low Grade Serous Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-06123; NCI-2019-06123 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10324 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10324 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Endometrial High Grade Endometrioid Adenocarcinoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube High Grade Serous Adenocarcinoma; Fallopian Tube Malignant Mixed Mesodermal (Mullerian) Tumor; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; FIGO Grade 1 Endometrial Endometrioid Adenocarcinoma; FIGO Grade 2 Endometrial Endometrioid Adenocarcinoma; Ovarian High Grade Serous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Undifferentiated Carcinoma; Platinum-Sensitive Ovarian Carcinoma; Primary Peritoneal Carcinosarcoma; Primary Peritoneal High Grade Serous Adenocarcinoma; Primary Peritoneal Transitional Cell Carcinoma; Primary Peritoneal Undifferentiated Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Low Grade Fallopian Tube Serous Adenocarcinoma; Recurrent Ovarian Carcinoma; Recurrent Ovarian Clear Cell Adenocarcinoma; Recurrent Ovarian Endometrioid Adenocarcinoma; Recurrent Ovarian Low Grade Serous Adenocarcinoma; Recurrent Ovarian Malignant Mixed Mesodermal (Mullerian) Tumor; Recurrent Ovarian Mucinous Adenocarcinoma; Recurrent Ovarian Transitional Cell Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Primary Peritoneal Low Grade Serous Adenocarcinoma
MeSH Terms: conditions — Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; liposomal doxorubicin; Doxorubicin; peposertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (peposertib, PLD) (Experimental): Patients receive peposertib PO BID on days 1-21, days 1-28, or days 1-7 (depending on dose level) and pegylated liposomal doxorubicin hydrochloride IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan or MRI during screening and every 8 weeks and after 6 months of study treatment, every 12 weeks. Patients undergo ECHO during screening and every 6 months. Starting in cycle 13, patients undergo ECHO or MUGA scan every 2 cycles. Additionally, patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Drug: Peposertib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Doxorubicin Liposomal; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
Drug: Peposertib — Given PO
  Other Names: 3-Pyridazinemethanol, alpha-(2-Chloro-4-fluoro-5-(7-(4-morpholinyl)-4-quinazolinyl)phenyl)-6-methoxy-, (alphaS)-; M 3814; M-3814; M3814; MSC 2490484A; MSC-2490484A; MSC2490484A; Nedisertib

SUMMARY:
This phase I trial studies the side effects and best dose of peposertib when given together with pegylated liposomal doxorubicin hydrochloride in treating patients with high or low grade ovarian cancer that has come back after a period of improvement (recurrent). Peposertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as pegylated liposomal doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving peposertib and pegylated liposomal doxorubicin hydrochloride may work better in treating patients with ovarian cancer compared to pegylated liposomal doxorubicin hydrochloride alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of peposertib (M3814) in combination with pegylated liposomal doxorubicin hydrochloride (PLD) and determine the recommended phase 2 dose (RP2D) of the combination in women with recurrent ovarian cancer.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate the pharmacokinetics of peposertib (M3814) when given in combination with PLD.

EXPLORATORY OBJECTIVE:

I. To correlate response to treatment (as defined by response rate and progression free survival) with PLD exposure (in area under the curve [AUC]) and PLD associated toxicities in women with recurrent high grade serous and low grade serous ovarian cancer treated in the expansion cohorts.

OUTLINE: This is a dose-escalation study of peposertib followed by a dose-expansion study.

Patients receive peposertib orally (PO) twice daily (BID) on days 1-21, days 1-28, or days 1-7 (depending on dose level) and pegylated liposomal doxorubicin hydrochloride intravenously (IV) on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients also undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) during screening and every 8 weeks throughout the study and after 6 months of study treatment, every 12 weeks. Patients undergo echocardiography (ECHO) during screening and every 6 months. Starting in cycle 13, patients undergo ECHO or multigated acquisition (MUGA) scan every 2 cycles. Additionally, patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* DOSE ESCALATION PHASE: Women with recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal cancer are eligible. This includes, but is not limited to, the following histologic types: serous adenocarcinoma (grade 1,2, or 3/ high grade or low grade), endometrioid adenocarcinoma, carcinosarcoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial adenocarcinoma, transitional cell carcinoma, or adenocarcinoma not otherwise specified

  * NOTE: Patients who have evidence of DDR deficiency /HRD are eligible if they are at the point in their disease course where they are appropriate candidates for single agent Doxil
* EXPANSION PHASE: The expansion phase will simultaneously accrue to 2 cohorts, low grade serous ovarian cancer (LGSOC) and high grade serous ovarian cancer (HGSOC)

  * Patients accrued to the LGSOC cohort will have recurrent or persistent low grade serous ovarian cancer or grade 1 serous ovarian cancer
  * Patients accrued to the HGSOC cohort will have recurrent or persistent high grade serous ovarian cancer
* Patients must have measurable disease by defined Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Prior therapy:

  * Patients must have received at least one prior line of platinum-based chemotherapy
  * Patients can have received an unlimited number of additional lines of chemotherapy, targeted therapy, biologic therapy, or hormonal therapy
  * Any prior therapy directed at the malignant tumor, including chemotherapy, biologic/targeted therapy, immunotherapy, or hormonal therapy must be discontinued at least 4 weeks, one cycle, or 5 half-lives (whichever is shortest) prior to study treatment initiation
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of peposertib (M3814) in combination with pegylated liposomal doxorubicin in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Patients with platinum-sensitive ovarian cancer are eligible for only the dose expansion phase if their provider feels that PLD would be an appropriate treatment option for them. Patients with platinum-sensitive ovarian cancer should also be offered any higher priority studies for which they are potentially eligible and/or platinum based chemotherapy or a PARP inhibitor if they are eligible for such therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Patients must have a cardiac ejection fraction >= the institutional lower limit of normal (LLN)
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Alkaline phosphatase =< 2.5 x institutional ULN
* Creatinine clearance > 30 ml/min
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression. The patient must be off steroids and clinically stable
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * The effects of peposertib (M3814) and liposomal doxorubicin on the developing human fetus are unknown and there is the potential for teratogenic or abortifacient effects. For this reason, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment, and for 6 months after completion of peposertib (M3814) administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with peposertib (M3814), breastfeeding should be discontinued if the mother is treated with peposertib (M3814)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* Archival formalin-fixed paraffin-embedded (FFPE) tissue collected within the past 36 months prior to registration must be available for submission for deoxyribonucleic acid (DNA)/ribonucleic acid (RNA) analysis

Exclusion Criteria:

* Patients are excluded from the dose-escalation phase of the study if they are eligible for any available therapies known to confer clinical benefit
* Inability to swallow and/or absorb oral medication (patients with a drainage peg are ineligible)
* Patients may not have received prior anthracyclines (doxorubicin or pegylated liposomal doxorubicin) for treatment of their ovarian cancer
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia, thyroid dysfunction, or neuropathy
* Patients who are receiving any other investigational agents within 28 days prior to start of treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to peposertib (M3814) or pegylated liposomal doxorubicin
* Patients who cannot discontinue concomitant medications or herbal supplements that potentially interact with peposertib (M3814)

  * The following categories of medications and herbal supplements must be discontinued prior to starting study treatment:

    * Strong inducers/inhibitors of CYP3A4/5, CYP2C9, and CYP2C19
    * Substrates with a narrow therapeutic index that are metabolized by CYP1A2, 2B6, 2C8, and 3A4/5
  * Use caution with other substrates of CYP3A4/5, CYP1A2, CYP2B6, CYP2C8 and substrates of P-gp, BCRP, OCT1, OAT3, OATP1B1, OATP1B3, MATE1, and MATE-2K with a narrow therapeutic index. Close monitoring is advised
  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. Patient Drug Interactions Handout and Wallet Card) should be provided to patients
* Patients who cannot discontinue concomitant proton-pump inhibitors (PPIs). Patients may confer with the study doctor to determine if such medications can be discontinued. These must be discontinued >= 5 days prior to study treatment. Patients do not need to discontinue calcium carbonate
* Patients receiving sorivudine or any chemically related analogues (such as brivudine) are excluded
* Patients who have received a live attenuated vaccine within 30 days of dosing with peposertib (M3814)
* Patients with uncontrolled intercurrent illness, including but not limited to ongoing or active infection
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because peposertib (M3814) is DNA-PK inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with peposertib (M3814), breastfeeding should be discontinued if the mother is treated with peposertib (M3814). These potential risks may also apply to other agents used in this study
* Patients with significant (uncontrolled) cardiac conduction abnormalities are excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  The descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 will be utilized for adverse event reporting.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameters of nedisertib | Up to 3 years
  Individual PK parameters will be estimated for maximum of concentration, area under the curve, T1/2, apparent clearance/oral bioavailability, and apparent volume using non-compartmental methods. The PK variables will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated for each dose level. Pharmacokinetic parameters will be reported descriptively for exploratory comparison with historical data. Samples from the expansion phase may also be analyzed for M3814 for the purpose of population-PK analyses.

OTHER OUTCOMES:
Tumor response | Within the first 10 months of treatment
  Tumor response will be defined according to Response Evaluation Criteria in Solid Tumors 1.1 and refers to the best overall response occurring.
Duration of response | From response documentation until progression of disease, assessed up to 3 years
Progression-free survival | From the beginning of the treatment until the progression date, death date, or the last radiological assessment without progressive disease, assessed up to 3 years
  Will be estimated using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel N Grisham, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (11):
- United States (11):
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT04092270/ICF_000.pdf